CLINICAL TRIAL: NCT03532464
Title: Randomized, Open-label, Multicenter Study of Azithromycin Compared With Doxycycline for Treating Anorectal Chlamydia Trachomatis Infection Concomitant to a Vaginal Infection
Brief Title: Azithromycin Compared With Doxycycline for Treating Anorectal Chlamydia Trachomatis Infection Concomitant to a Vaginal Infection
Acronym: CHLAZIDOXY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: USC EA 3671 Infections humaines à mycoplasmes et à chlamydiae (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2016/26
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Chlamydia Trachomatis Infection; Vaginal Infection; Anal Infection
Keywords: Chlamydia Trachomatis; Infection; Vaginal; Anal
MeSH Terms: conditions — Vaginitis; Infections | interventions — Azithromycin; Therapeutics; Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient treated by doxycycline (Experimental): The patients in the doxycycline group take one tablet of 100 mg twice a day for seven days.
  Antibiotics will be dispensed in their usual packaging with a clinical trial label.
  Interventions: Drug: doxycycline
- Patients treated by azithromycin (Active Comparator): The patients in the azithromycin group take 4 tablets of 250 mg in the morning as a single dose.
  Antibiotics will be dispensed in their usual packaging with a clinical trial label.
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: azithromycin — The route of administration is oral. It is administered at a dose of 1 g (4 tablets), as a single dose with or without food.
  Other Names: Treatment
  Arms: Patients treated by azithromycin
Drug: doxycycline — The patients in the doxycycline group take one tablet of 100 mg twice a day for seven days.
  Other Names: Treatment
  Arms: Patient treated by doxycycline

SUMMARY:
Chlamydia trachomatis is the most commonly reported bacterial sexually transmitted infection (STI), especially among young women. Up to 75% of C. trachomatis infected women are asymptomatic. If untreated, C. trachomatis infection can cause sequelae such as pelvic inflammatory disease, ectopic pregnancy and tubal factor infertility. C. trachomatis can also cause anorectal infections, which are typically asymptomatic. Among women with urogenital chlamydial infection, around 36-91% also had concurrent anorectal chlamydial. Notably, there was no association with anal intercourse in the studies that reported it. However, guidelines do not recommend routine anorectal testing, but restricted testing in people who are in high-risk groups, report anal sexual behavior, or have anal symptoms, i.e., on selective indications. This is in contrast to urogenital testing, which is a routine procedure in STI care services.

The anal transmission of C. trachomatis in women may occur by autoinoculation from the vagina due to the close proximity of the vagina and the anus. C. trachomatis could lead to a persistent infection in the lower gastrointestinal tract, suggesting the potential role of autoinoculation of cervical chlamydial infection from the rectal site. Such (repeat) urogenital infections could lead to reproductive tract morbidity. Recommended treatments for C. trachomatis infections are a single 1g dose of azithromycin or 100mg of doxycycline 2 times a day for 7 days. Although these two regimens are equivalent for urogenital infection, no study has compared the effectiveness of these two treatments on anorectal infection. If rectal C. trachomatis is a hidden reservoir influencing transmission rates, and considering the potential complications of cervical infections, providing further evidence of the need for effective rectal treatments among women is highly relevant.

DETAILED DESCRIPTION:
A possible reason for C. trachomatis detection after treatment may be transmission (self or another) or treatment failure. Whether antimicrobial treatment failure for C. trachomatis plays a role remains poorly understood. There is no evidence of antimicrobial resistance and testing for antimicrobial resistance for C. trachomatis is not routinely available. The hypothesis of transmission is most likely, especially as recontamination is very common among young people, either due to an untreated partner or a new partner. When these two conditions are ruled out, the hypothesis of autoinoculation from rectum to vagina is quite probable.

With regard to anorectal C. trachomatis infections, some studies concluded that azithromycin is a suboptimal treatment], while another study found doxycycline and azithromycin treatment to be equally effective. However, there are no robust studies that shows conclusive evidence relating to a suboptimal effect of any time of treatment or that prefers one treatment over the other.

The current study attempts to clarify the above question. The team propose to conduct the first open-label randomized controlled trial comparing the efficacy (measured as microbial cure) of a single 1g dose of azithromycin versus 100 mg of doxycycline twice daily for seven days for the treatment of anorectal C. trachomatis infection concurrent to urogenital infection in women. The experimental group will include women with C. trachomatis-positive vaginal and anorectal swabs treated with doxycycline twice daily for seven days with one tablet of 100 mg of doxycycline in the morning and evening. The control group will include women with C. trachomatis-positive vaginal and anorectal swabs treated with azithromycin consisting of four tablets of 250 mg of azithromycin in one intake.

The team made the hypothesis that the efficacy of azithromycin for anorectal infections may be lower than that of doxycycline, resulting in reinfections by autoinoculation from rectum to vagina. The expected result is that the number of women with a C. trachomatis-positive NAAT result in the anorectal swab will be significantly higher in the control group than in the experimental group after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* Negative β-hCG urinary assay and efficacious contraception for participant consulting in specialist centre
* Participant requesting an abortion at a pregnancy termination centre and efficacious contraception after abortion
* C. trachomatis-positive test for vaginal specimen using a Nucleic Acid Amplification Test (NAAT)
* Sexually active
* Consultation in one of the participating centers
* Agree to be contacted for follow-up
* Member or beneficiary of a social security system
* Free written informed consent signed by the participant and the investigator (no later than the inclusion day and before performing any examination required for the study)

Exclusion Criteria:

* Women who have symptoms suggesting pelvic inflammatory disease (PID)
* Receipt of an antibiotic with antichlamydial activity within 21 days before screening or between screening and enrollment
* Contraindications to tetracyclines, macrolides or ketolids (including allergy and treatment with colchicine, cisapride, ergot alkaloids and retinoids)
* Inability to swallow pills
* Refusal to participate in the study
* Objectives of the study not understood.
* Breast-feeding
* Patients with serious cardiac diseases: documented prolongation of the QT tract of the ECG, cardiac arrhythmias, advanced heart failure (classification New York Heart Association or NYHA >III)
* Patients treated with anticoagulants or drug with a definite potential of "Torsades de Pointe" or prolongation of the QT tract of the electrocardiogram
* Patients with severe liver diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A screening of vaginal C. trachomatis infection is performed among women consulting at a CeGIDD or at a termination pregnancy center before an abortion. C. trachomatis NAAT result will be available one week later, when the patient returns for consultation. In each participating center, a study site coordinator will screen all women with a C. trachomatis-positive vaginal swab and will verify eligibility criteria for inclusion in the study.
Enrollment: 460 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Nucleic Acid Amplification Assay result | 6 weeks
  C. trachomatis-positive NAAT result in anorectal specimens after treatment

SECONDARY OUTCOMES:
the number of women with an anorectal C. trachomatis infection concomitant to a vaginal infection | Day 1
  The prevalence of anorectal C. trachomatis infection concomitant to a vaginal infection is the number of women with an anorectal C. trachomatis infection divided by the total number of women included in the study
C. trachomatis genotype | Day 1
  The number of subjects for whom the same C. trachomatis genotype profile will be identified in the vaginal-positive and anorectal-positive specimens obtained on the day of inclusion (self-infection), and in the anorectal-positive specimen obtained six weeks after treatment initiation (persistence) and in the vaginal-positive specimen obtained four months after treatment (autoinoculation).
C. trachomatis genotype | 6 weeks
  The number of subjects for whom the same C. trachomatis genotype profile will be identified in the vaginal-positive and anorectal-positive specimens obtained on the day of inclusion (self-infection), and in the anorectal-positive specimen obtained six weeks after treatment initiation (persistence) and in the vaginal-positive specimen obtained four months after treatment (autoinoculation).
C. trachomatis genotype | 4 months
  The number of subjects for whom the same C. trachomatis genotype profile will be identified in the vaginal-positive and anorectal-positive specimens obtained on the day of inclusion (self-infection), and in the anorectal-positive specimen obtained six weeks after treatment initiation (persistence) and in the vaginal-positive specimen obtained four months after treatment (autoinoculation).

CONTACTS AND LOCATIONS:
Overall Officials: Bertille de Barbeyrac, MD, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CeGIDD - Marseille, Marseille, Marignane
  - CeGGID - Bordeaux, Bordeaux
  - CHU de Bordeaux, Bordeaux
  - CHU de Nantes, Nantes
  - Hôpital Hôtel Dieu, Paris
  - Hôpital de Roubaix, Roubaix
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rank RG, Yeruva L. Hidden in plain sight: chlamydial gastrointestinal infection and its relevance to persistence in human genital infection. Infect Immun. 2014 Apr;82(4):1362-71. doi: 10.1128/IAI.01244-13. Epub 2014 Jan 13. PMID 24421044
- [Result] Kong FY, Tabrizi SN, Fairley CK, Vodstrcil LA, Huston WM, Chen M, Bradshaw C, Hocking JS. The efficacy of azithromycin and doxycycline for the treatment of rectal chlamydia infection: a systematic review and meta-analysis. J Antimicrob Chemother. 2015 May;70(5):1290-7. doi: 10.1093/jac/dku574. Epub 2015 Jan 29. PMID 25637520
- [Result] Kong FY, Hocking JS. Treatment challenges for urogenital and anorectal Chlamydia trachomatis. BMC Infect Dis. 2015 Jul 29;15:293. doi: 10.1186/s12879-015-1030-9. PMID 26220080
- [Derived] Peuchant O, Lhomme E, Martinet P, Grob A, Baita D, Bernier C, Gibaud SA, Le Hen I, Le Naour E, Trignol-Viguier N, Lanotte P, Lefebvre P, Vachee A, Girard T, Loubinoux J, Bebear C, Ghezzoul B, Roussillon C, Kret M, de Barbeyrac B; CHLAZIDOXY Study Group. Doxycycline versus azithromycin for the treatment of anorectal Chlamydia trachomatis infection in women concurrent with vaginal infection (CHLAZIDOXY study): a multicentre, open-label, randomised, controlled, superiority trial. Lancet Infect Dis. 2022 Aug;22(8):1221-1230. doi: 10.1016/S1473-3099(22)00148-7. Epub 2022 May 9. PMID 35550262
- [Derived] Peuchant O, Lhomme E, Kret M, Ghezzoul B, Roussillon C, Bebear C, Perry F, de Barbeyrac B; and the Chlazidoxy study group. Randomized, open-label, multicenter study of azithromycin compared with doxycycline for treating anorectal Chlamydia trachomatis infection concomitant to a vaginal infection (CHLAZIDOXY study). Medicine (Baltimore). 2019 Feb;98(7):e14572. doi: 10.1097/MD.0000000000014572. PMID 30762806